CLINICAL TRIAL: NCT05246839
Title: Informed Choice Intervention for Colorectal Cancer Screening: Compass
Brief Title: Informed Choice - Compass
Status: Terminated | Type: Observational
Why Stopped: Business decision to terminate the study early. Primary endpoint will not be assessed.
Sponsor: Exact Sciences Corporation (Industry)
Collaborators: Mayo Clinic (Other); University of Utah (Other); American Cancer Society, Inc. (Other); F!ght Colorectal Cancer (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019-02
Record Dates: First submitted 2022-01-24; First posted 2022-02-18 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: CRC Screening; Colonoscopy; FIT; Cologuard; Screening Modality; Survey; Video; sDNA-FIT
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm 1 - Usual Care (No Video): Participant will receive the usual care pertaining to colorectal cancer (CRC) screening according to their respective clinical site and will not view either of the study videos.
- Arm 2 - Brief Video: Participant will watch a video pertaining to the importance of CRC screening.
  Interventions: Behavioral: Brief Video
- Arm 3 - Brief Video Plus: Participant will watch the same video as described in Arm 2, immediately followed by a second video pertaining to 3 CRC screening modalities: colonoscopy, FIT, and Cologuard.
  Interventions: Behavioral: Brief Video Plus

INTERVENTIONS:
Behavioral: Brief Video — Videos about colorectal cancer screening.
  Groups: Arm 2 - Brief Video
Behavioral: Brief Video Plus — Videos about colorectal cancer screening and modalities.
  Groups: Arm 3 - Brief Video Plus

SUMMARY:
The primary objective of this study is to evaluate the impact of a theoretically grounded video that includes information about CRC screening modality choices on CRC screening rates and time adherent to CRC guidelines. The results will not be posted because the study terminated early and the primary endpoint was not analyzed.

DETAILED DESCRIPTION:
Participants 45 to 70 years of age, scheduled for a primary care (index) appointment, at average risk for colorectal cancer (CRC), and due for CRC screening will be enrolled in the study. Participants will be randomized to one of three intervention arms: no video (arm 1), brief CRC screening video (arm 2), or enhanced CRC screening video (arm 3). Participants in all intervention arms will complete surveys regarding intention to screen for CRC and preference for screening modality prior to viewing the video, after the video, and after their index appointment. Participants will be surveyed, and medical information collected, for 1 year after randomization to assess adherence to CRC screening and CRC screening outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 45 to 70 years of age, inclusive.
2. Participant presents for a primary care appointment.
3. Participant understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information (PHI) to the study Investigator.
4. Participant has never been screened for CRC.

Exclusion Criteria:

1. Participant has symptoms or signs that require immediate, or near-term referral for diagnostic or therapeutic colonoscopy.
2. Participant is due for CRC screening within three months and is already scheduled for colonoscopy.
3. Participant has a personal history of CRC or colonic adenomatous or sessile serrated polyps.
4. Participant has a personal history of inflammatory bowel disease.
5. Participant has a family history of CRC in at least one first- or second-degree relative diagnosed prior to age 60 and/or at least 2 first-degree relatives diagnosed with CRC at any age.
6. Participant has a personal diagnosis or family history of any of the following conditions:

   1. Familial adenomatous polyposis (also referred to as "FAP", including attenuated FAP and Gardner's syndrome),
   2. Hereditary non-polyposis CRC syndrome (also referred to as "HNPCC" or "Lynch Syndrome"),
   3. Other hereditary cancer syndromes including, but are not limited to Peutz-Jeghers Syndrome, MYH-Associated Polyposis (MAP), Turcot's (or Crail's) Syndrome, Cowden's Syndrome, Juvenile Polyposis, Neurofibromatosis, or Familial Hyperplastic Polyposis.
7. Participant has a diagnosis of Cronkhite-Canada Syndrome.
8. Participant is current with CRC screening, including gFOBT or FIT within the preceding 12 months, Cologuard within the preceding 3 years, flexible sigmoidoscopy or CT colonography within the preceding 5 years, or colonoscopy within the preceding 10 years. Participants can be enrolled up to 3 months prior to screening due date.
9. Participant has any condition that in the opinion of the Investigators should preclude participation in the study, including comorbid illnesses precluding endoscopic evaluation or that limit life expectancy to less than 10 years.

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be 45 to 70 years of age, inclusive, who are scheduled for a primary care appointment, at average risk for colorectal cancer (CRC), and due for CRC screening. The study will enroll approximately 1,851 subjects.
Sampling Method: Probability Sample
Enrollment: 1823 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Impact of Brief Videos | 1 year
  To evaluate the impact of a theoretically grounded video that includes information about CRC screening modality choices (colonoscopy, FIT, and Cologuard) on CRC screening rates and the proportion of time adherent to CRC guidelines.

SECONDARY OUTCOMES:
Participant Screening Preferences | 1 year
  To examine initial mode preferences between participants viewing a theoretically grounded video that includes information about CRC screening modality choices (colonoscopy, FIT, and Cologuard) compared to those receiving only a brief informational video about CRC screening or receiving only usual care.

OTHER OUTCOMES:
Exploratory Objective- Participant | 1 year
  Evaluate participant knowledge, attitudes, and intentions related to CRC screening and assess personal and environmental factors associated with screening intentions and completion by modality.
Exploratory Objective- Provider | 1 year
  Characterize provider, system, and site-level factors associated with CRC screening rates and use of various screening modalities at different times throughout the intervention (prior to and after recruitment is completed).

CONTACTS AND LOCATIONS:
Overall Officials: Joan M. Griffin, PhD, Principal Investigator — Mayo Clinic College of Medicine; John Inadomi, MD, Principal Investigator — University of Utah; Charles R. Rogers, PhD, Principal Investigator — Rogers Solutions Group
Locations (39):
- United States (39):
  - Absolute Clinical Research, Phoenix, Arizona
  - Biopharma Informatic, Los Angeles, California
  - Saviers Medical Group, Port Hueneme, California
  - Skylight Health Group, Aurora, Colorado
  - Skylight Health Group, Jacksonville, Florida
  - I.V.A.M Clinical & Investigational Center, Miami, Florida
  - ITB Research, Miami, Florida
  - Emerald Coast OBGYN, Panama City, Florida
  - ClinCept, LLC, Columbus, Georgia
  - Pivotal Clinical Research & Associates, LLC, Marietta, Georgia
  - Herman Clinical Research, LLC, Suwanee, Georgia
  - Sheridan Medical Center, S.C, Chicago, Illinois
  - Ascension DePaul Community Services of New Orleans, New Orleans, Louisiana
  - Annapolis Internal Medicine, Annapolis, Maryland
  - Advanced Primary and Geriatric Care, Rockville, Maryland
  - Valley Ob-Gyn Clinic, PC, Saginaw, Michigan
  - St. Louis Medical Professionals, St Louis, Missouri
  - Barrett Clinic, La Vista, Nebraska
  - Alliance Community Healthcare, INC, Jersey City, New Jersey
  - North Hudson Community Action Corporation, Union City, New Jersey
  - Ellipsis Research Group, LLC, Brooklyn, New York
  - Niagara Falls Memorial Medical Center, Niagara Falls, New York
  - Laurelton Heart Specialist PC, Rosedale, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - Hightower Clinical OKC, Oklahoma City, Oklahoma
  - Skylight Health, Harrisburg, Pennsylvania
  - Mercado Medical Practice, Philadelphia, Pennsylvania
  - Pottstown Medical Specialists Inc, Pottstown, Pennsylvania
  - Center for Medical Research, LLC, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - SPICA Clinical Research, Columbia, South Carolina
  - The Jackson Clinic, PA, Jackson, Tennessee
  - Clear Brook Medical Associates, Houston, Texas
  - BioPharma Informatic, Pharr, Texas
  - Valena Medical Research, Spring, Texas
  - A & U Family Medicine, Sugarland, Texas
  - Ogden Clinic - Mountain View, Pleasant View, Utah
  - Ogden Clinic - Grand View, Roy, Utah
  - South Ogden Family Medicine, South Ogden, Utah

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in publications of the study may be shared after deidentification. This may include text, tables, figures, and appendices. The study protocol, statistical analysis plan (when applicable), informed consent form (when applicable), and clinical study report (when applicable) may also be shared. Data will be available from 2 years and ending 4 years after publication. Data may be shared with researchers who provide a methodologically sound proposal to achieve the aims outlined in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: Proposals for access to data should be directed to clinicaltrials@exactsciences.com. To gain access, data requestors will need to provide a methodologically sound proposal and sign a data access agreement. Researchers are required to obtain necessary IRB/EC approvals or waivers as applicable to conduct research. Data will be available between 2 and 4 years after publication through the Sponsor.
  For IPD related to Exact Sciences clinical studies, the Clinical Affairs department will include the policy description and access criteria described above with study-specific postings on clinicaltrials.gov.

REFERENCES:
- [Derived] Griffin JM, Finney Rutten LJ, Zhu X, Feng Z, Rogers CR, Marsh TL, Inadomi JM. The COMPASS study: A prospective, randomized, multi-center trial testing the impact of a clinic-based intervention informing patients of colorectal cancer screening options on screening completion. Contemp Clin Trials. 2022 Aug;119:106852. doi: 10.1016/j.cct.2022.106852. Epub 2022 Jul 13. PMID 35842109